CLINICAL TRIAL: NCT03040765
Title: Denosumab Versus Zoledronic Acid for Patients With Beta-Thalassemia Major-Induced Osteoporosis
Brief Title: Denosumab Versus Zoledronic Acid in Thalassemia-Induced Osteoporosis
Acronym: DOHA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: failed to recruit eligible subjects
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16441/16
Record Dates: First submitted 2017-01-22; First posted 2017-02-02 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-05

CONDITIONS: Thalassemia Majors (Beta-Thalassemia Major); Osteoporosis
Keywords: Osteoporosis; Beta-Thalassemia Major; Denosumab; Zoledronic Acid
MeSH Terms: conditions — beta-Thalassemia; Osteoporosis | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab (Active Comparator): Denosumab 60 MG/ML Prefilled Syringe
  Denosumab Dose: 60 milligrams, subcutaneous injection, every 6 months (twice a year)
  Interventions: Drug: Denosumab 60 MG/ML Prefilled Syringe
- Zoledronic Acid (Active Comparator): Zoledronic Acid 5Mg/Bag 100Ml Inj
  Zoledronic acid will be 5 milligrams, Intravenous injection, once a year
  Interventions: Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj

INTERVENTIONS:
Drug: Denosumab 60 MG/ML Prefilled Syringe — Denosumab 60 MG/ML will be administered to 20 patients with b-thalassemia major
  Other Names: Prolia
  Arms: Denosumab
Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj — Zoledronic Acid 5Mg/Bag 100Ml Inj will be administered to 20 patients with b-thalassemia major
  Other Names: Aclasta
  Arms: Zoledronic Acid

SUMMARY:
This study is to compare the two medications Denosumab and Zoledronic Acid For Patients With Beta Thalassemia Major Induced Osteoporosis. Patients with B-thalassemia major induce osteoporosis will undergo baseline assessment of the bone densitometry by Dual-energy X-ray absorptiometry scan as a standard of care by the radiology department, then a blood test for bone specific Alkaline phosphatase and type-1 Carboxy Telopeptide will be measured by the chemistry lab.

Patients with B-Thalassemia Major induced osteoporosis, who are 18 years of age or more and willing to participate in the study will be enrolled after consenting by the primary investigator in hematology outpatient clinic. Patients with osteoporosis will receive one of the two medications, at the end of the year Dual-energy X-ray absorptiometry scan will be done to compare the response of the two medications. The potential risks include the drug-related side effects

DETAILED DESCRIPTION:
Despite the significant improvements in the therapeutic management of beta thalassemia major (BTM) over the past few decades, osteoporosis is still a common finding, even in optimally treated patients. The relationships between bone mineral densities (BMD) and several clinical characteristics or hematological markers have been described. Chronic anemia, bone marrow expansion due to ineffective erythropoiesis, iron toxicity, calcium and zinc deficiencies, low vitamin D levels and endocrine complications have been suggested to contribute to the etiology of bone diseases in BTM. Nevertheless, the complex etiological mechanisms of this heterogeneous osteopathy remain incompletely clarified. A complex mechanism controls bone remodeling in human. This mechanism includes the receptor activator of nuclear factor kappa B ligand (RANKL), its natural receptor (RANK) and osteoprotegerin (OPG). The RANK/RANKL pathway is an essential to promote osteoclast formation and activation and prolongs osteoclast survival.

OPG acts as a decoy receptor for RANKL and prevents its interaction with RANK thereby inhibiting osteoclast formation, function, and survival. Alteration of the RANK/RANKL/OPG system for increased osteoclastic activity and enhanced osteoblastic dysfunction is proposed as an important mechanism in the etiology of osteoporosis in BTM. Hypogonadism, a common finding in BTM, is associated with enhanced RANKL activity. The sex steroid hormones, androgen, and estrogens, via their respective nuclear receptors, regulate BMD in humans and mice. Testosterone is likely to have direct and indirect inhibitory effects on human osteoclast formation and bone resorption. Animal model and cell culture studies suggest a direct inhibitory effect of androgens on the OPG/RANKL cytokines system. In human osteoblastic cells, testosterone and 5-dihydrotestosterone mediate an androgen receptor-induced specific inhibition of OPG messenger ribonucleic acid (mRNA) expression. Androgens have also been shown to block RANKL-induced osteoclastic formation while RANKL expression was found to be up-regulated in osteoblastic cells from androgen receptor-deficient mice. The effect of oestradiol (E2) on osteoclast precursors and osteoclasts seems to be mediated by osteoblastic cells. Inhibitory effect of E2 is associated with the stimulated secretion of OPG by osteoblasts. Previous studies have focused on the characteristics of thalassemic patients with osteoporosis and their response to therapy with bisphosphonate. Because RANK-RANKL and OPG play a significant role in bone resorption and seem to be the principal implicated mechanism for the development of osteoporosis in BTM, we will conduct this prospective study to evaluate the anti-RANKL denosumab versus zoledronic acid on TM-induced osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Age 18 years old or older
* Eastern Cooperative Oncology Group Performance Status less than or equal 2

Exclusion Criteria:

* Age less than 18 years old
* Not willing to participate in the study
* Vulnerable subjects or Eastern Cooperative Oncology Group Performance Status 3 or 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with a 50 percent or greater reduction in type-1 collagen carboxy telopeptide from the baseline | 12 months
  Number of patients with a 50 percent or greater reduction in type-1 collagen carboxy telopeptide from the baseline

SECONDARY OUTCOMES:
Number of patients with a 50 percent or greater improvement in Dual-energy X-ray absorptiometry scan from the baseline | 12 months
  Number of patients with a 50 percent or greater improvement in Dual-energy X-ray absorptiometry scan from the baseline
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Yassin, Principal Investigator — Hamad Medical Corporation
Locations (1):
- National Center for Cancer Care & Research (NCCCR), Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baldini M, Forti S, Marcon A, Ulivieri FM, Orsatti A, Tampieri B, Airaghi L, Zanaboni L, Cappellini MD. Endocrine and bone disease in appropriately treated adult patients with beta-thalassemia major. Ann Hematol. 2010 Dec;89(12):1207-13. doi: 10.1007/s00277-010-1007-0. Epub 2010 Jun 26. PMID 20582415
- [Background] Scacchi M, Danesi L, Cattaneo A, Valassi E, Pecori Giraldi F, Argento C, D'Angelo E, Mirra N, Carnelli V, Zanaboni L, Tampieri B, Cappellini MD, Cavagnini F. Bone demineralization in adult thalassaemic patients: contribution of GH and IGF-I at different skeletal sites. Clin Endocrinol (Oxf). 2008 Aug;69(2):202-7. doi: 10.1111/j.1365-2265.2008.03191.x. Epub 2008 Jan 21. PMID 18221395
- [Background] Kyriakou A, Savva SC, Savvides I, Pangalou E, Ioannou YS, Christou S, Skordis N. Gender differences in the prevalence and severity of bone disease in thalassaemia. Pediatr Endocrinol Rev. 2008 Oct;6 Suppl 1:116-22. PMID 19337164
- [Background] Voskaridou E, Terpos E. Pathogenesis and management of osteoporosis in thalassemia. Pediatr Endocrinol Rev. 2008 Oct;6 Suppl 1:86-93. PMID 19337161
- [Background] Pietrapertosa AC, Minenna G, Colella SM, Santeramo TM, Renni R, D'Amore M. Osteoprotegerin and RANKL in the pathogenesis of osteoporosis in patients with thalassaemia major. Panminerva Med. 2009 Mar;51(1):17-23. PMID 19352306
- [Background] Mahachoklertwattana P, Pootrakul P, Chuansumrit A, Choubtum L, Sriphrapradang A, Sirisriro R, Rajatanavin R. Association between bone mineral density and erythropoiesis in Thai children and adolescents with thalassemia syndromes. J Bone Miner Metab. 2006;24(2):146-52. doi: 10.1007/s00774-005-0661-0. PMID 16502122
- [Background] Aslan I, Canatan D, Balta N, Kacar G, Dorak C, Ozsancak A, Oguz N, Cosan R. Bone mineral density in thalassemia major patients from antalya, Turkey. Int J Endocrinol. 2012;2012:573298. doi: 10.1155/2012/573298. Epub 2012 Jun 20. PMID 22778734
- [Background] Pincelli AI, Masera N, Tavecchia L, Perotti M, Perra S, Mariani R, Piperno A, Mancia G, Grassi G, Masera G. GH deficiency in adult B-thalassemia major patients and its relationship with IGF-1 production. Pediatr Endocrinol Rev. 2011 Mar;8 Suppl 2:284-9. PMID 21705979
- [Background] Pirinccioglu AG, Akpolat V, Koksal O, Haspolat K, Soker M. Bone mineral density in children with beta-thalassemia major in Diyarbakir. Bone. 2011 Oct;49(4):819-23. doi: 10.1016/j.bone.2011.07.014. Epub 2011 Jul 23. PMID 21798385
- [Background] Skordis N, Ioannou YS, Kyriakou A, Savva SC, Efstathiou E, Savvides I, Christou S. Effect of bisphosphonate treatment on bone mineral density in patients with thalassaemia major. Pediatr Endocrinol Rev. 2008 Oct;6 Suppl 1:144-8. PMID 19337169
- [Background] Soliman AT, El Banna N, Abdel Fattah M, ElZalabani MM, Ansari BM. Bone mineral density in prepubertal children with beta-thalassemia: correlation with growth and hormonal data. Metabolism. 1998 May;47(5):541-8. doi: 10.1016/s0026-0495(98)90237-2. PMID 9591744
- [Background] Mahachoklertwattana P, Chuansumrit A, Sirisriro R, Choubtum L, Sriphrapradang A, Rajatanavin R. Bone mineral density, biochemical and hormonal profiles in suboptimally treated children and adolescents with beta-thalassaemia disease. Clin Endocrinol (Oxf). 2003 Mar;58(3):273-9. doi: 10.1046/j.1365-2265.2003.01707.x. PMID 12608931
- [Background] Boyce BF, Xing L. Functions of RANKL/RANK/OPG in bone modeling and remodeling. Arch Biochem Biophys. 2008 May 15;473(2):139-46. doi: 10.1016/j.abb.2008.03.018. Epub 2008 Mar 25. PMID 18395508
- [Background] Kearns AE, Khosla S, Kostenuik PJ. Receptor activator of nuclear factor kappaB ligand and osteoprotegerin regulation of bone remodeling in health and disease. Endocr Rev. 2008 Apr;29(2):155-92. doi: 10.1210/er.2007-0014. Epub 2007 Dec 5. PMID 18057140
- [Background] Pepene CE, Crisan N, Coman I. Elevated serum receptor activator of nuclear factor kappa B ligand and osteoprotegerin levels in late-onset male hypogonadism. Clin Invest Med. 2011 Aug 1;34(4):E232. doi: 10.25011/cim.v34i4.15365. PMID 21810381
- [Background] Michael H, Harkonen PL, Vaananen HK, Hentunen TA. Estrogen and testosterone use different cellular pathways to inhibit osteoclastogenesis and bone resorption. J Bone Miner Res. 2005 Dec;20(12):2224-32. doi: 10.1359/JBMR.050803. Epub 2005 Aug 1. PMID 16294275
- [Background] Hofbauer LC, Hicok KC, Chen D, Khosla S. Regulation of osteoprotegerin production by androgens and anti-androgens in human osteoblastic lineage cells. Eur J Endocrinol. 2002 Aug;147(2):269-73. doi: 10.1530/eje.0.1470269. PMID 12153751
- [Background] Grundt A, Grafe IA, Liegibel U, Sommer U, Nawroth P, Kasperk C. Direct effects of osteoprotegerin on human bone cell metabolism. Biochem Biophys Res Commun. 2009 Nov 20;389(3):550-5. doi: 10.1016/j.bbrc.2009.09.026. Epub 2009 Sep 11. PMID 19748486
- [Background] Huber DM, Bendixen AC, Pathrose P, Srivastava S, Dienger KM, Shevde NK, Pike JW. Androgens suppress osteoclast formation induced by RANKL and macrophage-colony stimulating factor. Endocrinology. 2001 Sep;142(9):3800-8. doi: 10.1210/endo.142.9.8402. PMID 11517156
- [Background] Kawano H, Sato T, Yamada T, Matsumoto T, Sekine K, Watanabe T, Nakamura T, Fukuda T, Yoshimura K, Yoshizawa T, Aihara K, Yamamoto Y, Nakamichi Y, Metzger D, Chambon P, Nakamura K, Kawaguchi H, Kato S. Suppressive function of androgen receptor in bone resorption. Proc Natl Acad Sci U S A. 2003 Aug 5;100(16):9416-21. doi: 10.1073/pnas.1533500100. Epub 2003 Jul 18. PMID 12872002
- [Background] Gorny G, Shaw A, Oursler MJ. IL-6, LIF, and TNF-alpha regulation of GM-CSF inhibition of osteoclastogenesis in vitro. Exp Cell Res. 2004 Mar 10;294(1):149-58. doi: 10.1016/j.yexcr.2003.11.009. PMID 14980510